CLINICAL TRIAL: NCT02641158
Title: CTN 0064: Assessing Long-term CTN 0049 Outcomes, HCV Prevalence and Progression Along the HCV Care Continuum Among HIV/HCV Co-infected Substance Users in the U.S.
Brief Title: Assessing Long-term CTN 0049 Outcomes, HCV Prevalence and Progression Along the HCV Care Continuum Among HIV/HCV Co-infected Substance Users in the U.S.
Acronym: CTN 0064
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Jackson Health System (Other); Grady Memorial Hospital (Other); St. Luke's-Roosevelt Hospital Center (Other); University of Texas (Other); Johns Hopkins University (Other); University Hospital Birmingham (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); University of Pittsburgh Medical Center (Other); Hahnemann University Hospital (Other); Cook County Health (Other Government); Boston University (Other); Weill Medical College of Cornell University (Other); Icahn School of Medicine at Mount Sinai (Other); The Emmes Company, LLC (Industry); University of Miami (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Lisa Metsch, Stephen Smith Professor and Chair of Sociomedical Sciences Department, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAP8757; U10DA013720 (NIH)
Record Dates: First submitted 2015-12-13; First posted 2015-12-29 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C; HIV; AIDS; Substance Use
Keywords: HIV; Hepatitis C; Substance users; Drug users
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Drug Misuse | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Other)
  Interventions: Other: Control Group
- Care Facilitation Group (Experimental)
  Interventions: Behavioral: Care Facilitation Group

INTERVENTIONS:
Other: Control Group — After screening HCV antibody positive, participants will receive an appointment and reminder card to return for their HCV RNA results. If HCV RNA positive, study staff will attempt to make an appointment for the participant's next step in the HCV continuum. If a participant attends the "next step" visit, the participant would be subject to whatever is the local standard of care at that clinic/agency from that point forward.
  Arms: Control Group
Behavioral: Care Facilitation Group — The same will occur for intervention participants, yet an HCV care facilitator will motivate them to return for their HCV RNA results; appointment reminders will be made prior to the "next step" visit; follow-up contact will be made for missed appointments; and the HCV care facilitator will coordinate and link the participant to available community resources (e.g., mental health, housing agencies) by scheduling appointments, arranging transportation, and helping to complete any clinic registration (or other) paperwork that agencies may require to access services.
  Arms: Care Facilitation Group

SUMMARY:
Primary Objective: This study will evaluate the effectiveness of an HCV Care Facilitation intervention in moving HIV/HCV co-infected substance users forward along the HCV care continuum (compared with a Control group).

Primary Hypothesis: The number of steps achieved along the HCV care continuum will differ between the two study groups over the 14-month follow-up period.

Secondary Objectives:

Component 1 (Long-term CTN 0049 follow-up):

Using the CTN 0064 baseline data (self-report, medical record abstraction and biological data), the following CTN 0049 primary and secondary outcomes in participants who consented to the CTN 0064 protocol will be re-analyzed to evaluate latent and/or enduring effects of the CTN 0049 interventions:

1. HIV virological suppression
2. HIV primary care visit attendance
3. All-cause mortality

DETAILED DESCRIPTION:
The CTN 0064 study leverages the existing research infrastructure and cohort of the CTN 0049 (NCT01612169) randomized, controlled trial (RCT). CTN 0049 ("Project HOPE -- Hospital Visit as Opportunity for Prevention and Engagement for HIV-Infected Drug Users") is a three-group RCT that evaluated the most effective strategy to achieve HIV virologic suppression among HIV-infected substance users who were recruited from hospital settings. Between July 2012 and January 2014, a total of 801 HIV-infected hospitalized patients were recruited from 11 participating sites throughout the U.S. and randomized to one of the following three groups: 1) Patient Navigator intervention, 2) Patient Navigator plus Contingency Management intervention, and 3) Treatment as Usual. All CTN 0049 participants provided informed consent and completed baseline computer assisted personal interviews or CAPI (computer assisted personal interview: focusing on drug use, mental health, demographics and socio-economic factors, HIV care and drug treatment history) and blood draws (for HIV viral load and CD4 count). The two intervention groups received up to 11 patient navigation sessions over a 6-month period to actively assist participants in linking to HIV primary care and substance use treatment. Participants in all three groups completed follow-up assessments consisting of CAPI, blood draws, urine collection and breath analysis at approximately 6 and 12 months post-randomization. Medical records were reviewed to document receipt of HIV care and treatment during the study period. CTN 0064 will leverage the CTN 0049 research infrastructure and cohort by utilizing the 11 participating CTN 0049 research teams to recruit their randomized participants into the CTN 0064 study.

CTN 0064 has two main components: Component 1 is the baseline assessment for CTN 0064. It will also serve as a long-term follow-up assessment for CTN 0049 for those who consent to participate in CTN 0064. Participants whose HCV antibody test result is positive in this baseline assessment will be invited to enroll in Component 2. Component 2 is an RCT that will assess the effectiveness of a Care Facilitation intervention (compared to Control) in moving HIV/HCV co-infected substance users forward along the HCV care continuum. The study's primary objective is based on Component 2 and will be operationalized as movement through a series of (potentially non-sequential) pre-defined, clinical steps along the HCV care continuum (including the ultimate step, sustained virologic response to treatment at 12 weeks post treatment completion [SVR12]) (AASLD/IDSA/IAS-USA). Secondary objectives will be to assess: 1) success at each step in the HCV care continuum, 2) engagement in HIV care and substance use treatment, and 3) HIV viral suppression as well as 4) to examine other long-term outcomes of the CTN 0049 cohort.

All adults who were randomized into the CTN 0049 study and who provided consent to be contacted about future studies (hereafter, referred to as the "CTN 0049 cohort") will be invited to enroll in the CTN 0064 study. All participants will provide informed consent and complete Component 1, consisting of: 1) a computer assisted personal interview or CAPI (capturing history of HIV care, HCV testing and care, substance use and substance use treatment; mental health; demographics; and socio-economic factors), 2) HCV antibody screening via rapid HCV test (and, if HCV antibody positive, HCV RNA testing via venipuncture), 3) associated pre-/post-HCV test information and counseling, 4) blood specimen collection via venipuncture, and 5) drug/alcohol toxicology screening (via urine evaluation). The blood specimens of all participants will be assessed for HIV viral load and CD4 count. The blood specimens for the subset of participants who screen as HCV antibody positive will be assessed for HCV RNA to determine if their HCV infection is active.

Participants who screen as HCV antibody positive will be randomized into Component 2 and assigned to one of two groups: 1) HCV Care Facilitation intervention or 2) Control. The Care Facilitation intervention group will receive up to 12 sessions during a 6-month intervention period. Follow-up visits with both groups will be conducted at approximately 6 and 12 months post-randomization. These visits will consist of CAPI, blood specimen collection, and drug/alcohol toxicology screening. Medical records will be reviewed to document HCV testing, receipt and use of HCV clinical evaluation, care and treatment (as applicable); and HIV care and treatment before and during the study period.

ELIGIBILITY:
Inclusion Criteria:

By virtue of participating individuals being recruited from the CTN-0049 cohort, they will be:

1. HIV-infected and
2. 18 years of age or older
3. Be able to communicate in English

   Additionally, to be eligible for Component 1 they must:
4. provide informed consent, which includes being willing to provide sufficient locator information and to be tested for anti-HCV antibodies and, if antibody positive, tested for active HCV infection
5. sign a HIPAA form / medical record release form to facilitate medical record abstraction

   Finally, to continue on to Component 2, they must:
6. provide sufficient locator information
7. report living in the vicinity and being able to return for follow-up visits
8. complete the baseline assessments
9. complete the blood draw
10. test as HCV antibody positive via study Component 1 and,
11. agree to be randomized in Component 2

Exclusion Criteria:

Individuals will be excluded from participation if they:

1. have significant cognitive or developmental impairment
2. are terminated via Site Principal Investigator decision/discretion with agreement from study Lead Investigator
3. are currently in jail, prison or any inpatient overnight facility as required by court of law or have a pending legal action which may prevent an individual from completing the study

   Additionally, individuals may participate in Component 1, but will be excluded from Component 2 if they:
4. are currently on HCV therapy/medications at baseline
5. have completed a course of HCV medications in the last 12 weeks based on self-report.

It should be noted that pregnancy is not an exclusion criterion. Therefore, sites may enroll pregnant women and/or follow-up with already enrolled women who become pregnant after enrollment in the study provided that they have local IRB approval to do so.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2015-12; Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Forward movement along the HCV care continuum assessed as the difference between the number of steps completed pre- and post-randomization (among Component 2 participants) | 14 months post-randomization (this is the outside window for the 12-month follow-up visit)
  The primary outcome is a count variable: total # of completed steps along the HCV care continuum by 14 months post-randomization (this is the outside window for the 12-month follow-up visit) minus the total number of steps completed within 12 months prior to baseline. Participants' final step on the HCV care continuum will be assessed the last time they are observed in medical records within the 14-month-long follow-up period. Because the entire sample has HIV, we include 2 HIV-related steps:
  1. Receipt of HCV RNA result -- result received within 3 months of baseline
  2. HIV primary care visit -- completion of 1 visit with an HIV primary care provider
  3. Initiated HIV ART
  4. HCV evaluation
  5. HCV treatment offered and declined or prescription process initiated
  6. HCV treatment initiated
  7. Course of HCV treatment completed
  8. SVR12 (sustained virologic response) achieved at 12 or more weeks after treatment completion

SECONDARY OUTCOMES:
HIV viral suppression | Assessed at the CTN 0064 baseline visit
  Suppression binary defined as viral load <=200 copies/ml (yes) vs. viral load >200 copies/ml or all-cause mortality (no)
HIV care visit attendance | Assessed in the 6-month time period before the CTN 0064 baseline visit
All-cause mortality | Time period will vary by participant between 9 months and 4 years depending when they were randomized into CTN 0049 and when they complete the CTN 0064 baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R. Metsch, PhD, Principal Investigator — Columbia University; Carlos del Rio, MD, Principal Investigator — Emory University; Daniel J. Feaster, PhD, Principal Investigator — University of Miami; Carmen Masson, PhD, Principal Investigator — University of California, San Francisco; David Perlman, MD, Principal Investigator — Mount Sinai Icahn School of Medicine; Lauren K. Gooden, PhD, Study Director — Columbia University
Locations (11):
- United States (11):
  - University Hospital at University of Alabama at Birmingham, Birmingham, Alabama
  - Los Angeles BioMedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Jackson Health System Adult HIV Outpatient Clinics / University of Miami, Miami, Florida
  - Grady Memorial Hospital / Ponce de Leon Center, Atlanta, Georgia
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Johns Hopkins Hospital / Moore Clinic, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Mount Sinai - St. Luke's Roosevelt Hospital Center, New York, New York
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian / Pittsburgh AIDS Center for Treatment, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Information about the study and the de-identified study data will be available at https://datashare.nida.nih.gov/ within 18 months of the date the data are locked, as per the procedures of the National Drug Abuse Treatment Clinical Trials Network.
Time Frame: Within 18 months.
Access Criteria: Information will be de-identified.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Derived] Gutkind S, Starbird LE, Murphy SM, Teixeira PA, Gooden LK, Matheson T, Feaster DJ, Jain MK, Masson CL, Perlman DC, Del Rio C, Metsch LR, Schackman BR. Cost of Hepatitis C care facilitation for HIV/Hepatitis C Co-infected people who use drugs. Drug Alcohol Depend. 2022 Mar 1;232:109265. doi: 10.1016/j.drugalcdep.2022.109265. Epub 2022 Jan 10. PMID 35042101
- [Derived] Metsch LR, Feaster DJ, Gooden LK, Masson C, Perlman DC, Jain MK, Matheson T, Nelson CM, Jacobs P, Tross S, Haynes L, Lucas GM, Colasanti JA, Rodriguez A, Drainoni ML, Osorio G, Nijhawan AE, Jacobson JM, Sullivan M, Metzger D, Vergara-Rodriguez P, Lubelchek R, Duan R, Batycki JN, Matthews AG, Munoz F, Jelstrom E, Mandler R, Del Rio C. Care Facilitation Advances Movement Along the Hepatitis C Care Continuum for Persons With Human Immunodeficiency Virus, Hepatitis C, and Substance Use: A Randomized Clinical Trial (CTN-0064). Open Forum Infect Dis. 2021 Jun 27;8(8):ofab334. doi: 10.1093/ofid/ofab334. eCollection 2021 Aug. PMID 34377726